CLINICAL TRIAL: NCT04400123
Title: A Single-centre, Single-dose, Randomized, Open-label and Two-cycle Crossover Bioequivalence Study of Famitinib Malate Capsules in Old and New Formulation on Healthy Chinese Subjects
Brief Title: A Bioequivalence Study of Famitinib Malate on Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: FMTN-I-103
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Healthy Adult Subjects
Keywords: Bioequivalence; Old formulation; New formulation

STUDY DESIGN:
Intervention Model Description: Treatment group TR Intervention: Drug: famitinib malate, new formulation; Intervention: Drug: famitinib malate, old formulation.
  Treatment group RT Intervention: Drug: famitinib malate, old formulation; Intervention: Drug: famitinib malate, new formulation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group TR (Experimental): Intervention: Drug: famitinib malate, new formulation; Intervention: Drug: famitinib malate, old formulation.
  Interventions: Drug: Famitinib malate
- Treatment group RT (Experimental): Intervention: Drug: famitinib malate, old formulation; Intervention: Drug: famitinib malate, new formulation.
  Interventions: Drug: Famitinib malate

INTERVENTIONS:
Drug: Famitinib malate — TR group:
  The first period，the subjects will be administrated with Famitinib malate in new formulation, then conduct blood collection within 192h; 14 days washout；The second period，the subjects will be administrated with Famitinib malate in old formulation, then conduct blood collection within 192h.
  RT group:
  The first period，the subjects will be administrated with Famitinib malate in old formulation, then conduct blood collection within 192h; 14 days washout；The second period，the subjects will be administrated with Famitinib malate in new formulation, then conduct blood collection within 192h.

SUMMARY:
The primary objective is to evaluate the bioequivalence of famitinib malate capsules in new and old formulations after oral dose under fasted condition on healthy Chinese subjects.

The secondary objective is to evaluate the safety after famitinib malate capsules oral dose on healthy Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects aged 18~45 (including 18 and 45 years old);
2. Body weight ≥ 50kg, body mass index (BMI) within the range of 19 ~ 26kg/m2 (including 19 and 26 kg/m2) (BMI= weight (kg)/height 2 (m2));
3. Consent to abstinence or take effective non-drug contraception measures during the study and for at least 3 months after the last drug administration.
4. The subjects were able to communicate well with the researchers, understand and comply with the requirements of this study, understand and sign the informed consent;

Exclusion Criteria:

1. Anyone who has suffered from any clinical serious disease such as the circulatory system, endocrine system, nervous system, digestive system, respiratory system, urogenital system, hematology, immunology, psychiatry and metabolic abnormalities, or any other disease which can affect the study results.
2. Those who have undergone surgery within 6 months before the trial, or plan to perform surgery during the study period;
3. Those who donated blood or suffered heavy blood loss (≥200 mL), received blood transfusions, or used blood products within 3 months before enrollment;
4. Have a history of allergies to drugs, food or other substances;
5. Have taken sedatives, sleeping pills or other addictive medicines within 1 year before the study; Those with positive results in urine drug abuse screening;
6. Those who have participated in any clinical trials and have taken study drugs within 3 months before the first administration;
7. Those who have taken any medicine within 4 weeks before the first administration (including prescription medicines, non-prescription medicines, Chinese herbal medicines, vitamins, calcium tablets and other food supplements);
8. Those who smoked more than 5 cigarettes per day within 3 months before the study and who could not stop using any tobacco products during the study;
9. Regular drinkers within 6 months before the test, that is, drinking more than 14 units of alcohol per week (1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine), and any alcohol-containing products cannot be stopped during the study Those who are positive for alcohol breath test;
10. Those with any abnormal result (clinically significant) of vital signs, physical examination, 12-lead electrocardiogram, chest radiograph, abdominal ultrasound, colour Doppler echocardiography, hematology, clinical chemistry, urinalysis and coagulation;
11. Hepatitis B virus surface antigen is positive, or hepatitis C virus antibody is positive, or treponema pallidum antibody is positive, or human immunodeficiency virus antibody is positive;
12. The subject refuses to stop any beverage or food containing methylxanthine, such as coffee, tea, cola, chocolate, etc., within 48 hours before the first dose until the end of the study; The subject refuses to stop any beverage or food containing grapefruit; Those who have special dietary requirements and cannot accept the unified diet;
13. Other factors of the subject that are not suitable for participating in the study judged by the investigators.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2020-07-18 (Actual); Study Completion 2020-07-18 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameter: Cmax | through study completion, an average of 30 days
  Peak plasma concentration （Cmax）
Pharmacokinetics parameter: AUC | through study completion, an average of 30 days
  Area under the plasma concentration versus time curve（AUC）

SECONDARY OUTCOMES:
Pharmacokinetics parameter: Tmax | through study completion, an average of 30 days
  Time of maximum observed concentration (Tmax)
Pharmacokinetics parameter: t1/2 | through study completion, an average of 30 days
  Half time (t1/2)
Pharmacokinetics parameter: λz | through study completion, an average of 30 days
  First order elimination rate constant (λz)
The number of participants with treatment-related adverse events assessed by CTCAE V5.0 | through study completion, an average of 30 days
  An adverse event is any untoward medical occurrence in the subjects or clinical study participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital Beijing, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided